CLINICAL TRIAL: NCT04496778
Title: The Beneficial Effect of Low Level Laser Therapy Combined With Nasal Irradiation on Cognitive Function and Quality of Life in Alzheimer Anemic Elderly Patients
Brief Title: Low Level Laser Therapy Impact on Cognitive Function and Quality of Life in Alzheimer Anemic Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ebtesam Nabil, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/0027772
Record Dates: First submitted 2020-07-27; First posted 2020-08-03 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer Disease; Cognitive Impairment, Mild
Keywords: low level laser; quality of life
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Low-Level Light Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low level laser plus exercise (Active Comparator): acupuncture low level laser combined with nasal laser irradiation in addition to aerobic exercise 3 times per week for 3 months
  Interventions: Device: low level laser therapy ( laser acupuncture combined with nasal laser irradiation); Other: aerobic exercise
- sham laser plus exercise (Placebo Comparator): placebo acupuncture low level laser combined with nasal laser irradiation in addition to aerobic exercise 3 times per week for 3 months
  Interventions: Device: low level laser therapy ( laser acupuncture combined with nasal laser irradiation); Other: aerobic exercise

INTERVENTIONS:
Device: low level laser therapy ( laser acupuncture combined with nasal laser irradiation) — Cold Laser Therapy Watch (Laser Watch- 650 nm) combines acupuncture and nasal cavity for external blood irradiation. Laser watch with 10 laser beams - is applied to the left wrist.
  Nasal Probe with 2 laser beams - is applied to the nose cavity
Other: aerobic exercise — 3 d/week for 45 to 60 minutes per session for 3 months. started by 40%-50% Heart Rate Reserve (determined by using a walking treadmill exercise test) during the first 6 weeks increasing gradually up to 50%-70% Heart Rate Reserve

SUMMARY:
Alzheimer's is a type of dementia that affects memory, thinking and behavior. Symptoms eventually grow severe enough to interfere with daily tasks. this study aimed to delay the deterioration of anemic elderly condition as memory affection interfere with daily life activities and social interaction

DETAILED DESCRIPTION:
Alzheimer's disease is the commonest cause of dementia and describes a clinical syndrome made up of three domains. First, a neuro-psychological domain encompassing those deficits of cognitive function such as amnesia (memory loss), aphasia (language disturbance), apraxia (the inability to carry out motor tasks despite intact motor functions) and agnosia (the inability to recognize people or objects despite intact sensory functions). Second, a group of psychiatric symptoms and behavioral disturbances, which have been termed neuro-psychiatric features, non-cognitive phenomena, or behavioral and psychological symptoms of dementia Alzheimer's disease is substantially increased among people aged 65 years or more, with a progressive decline in memory, thinking, language and learning capacity. Alzheimer's disease should be differentiated from normal age-related decline in cognitive function, which is more gradual and associated with less disability. Diabetes, hypertension, smoking, obesity, and dyslipidemia have all been found to increase risk as well a history of brain trauma, cerebrovascular disease, and vasculopathies.

Dementia affects approximately 5%-8% of individuals over age 65, 15%- 20% of individuals over age 75, and 25%-50% of individuals over age 85. Alzheimer disease is the most common dementia, accounting for 50%-75% of the total, with a greater proportion in the higher age ranges Dementia is expensive. The financial costs of managing Alzheimer's disease are enormous. The cost of illness is high in terms of both public and private resources. Families and caregivers who are required to provide care and patients affected by dementia also pay a high price in terms of their quality of life The primary goals of treatment are to maximize the patient's ability to function in daily life, maintain quality of life, slow the progression of symptoms, and treat depression or disruptive behaviors Low level laser therapy is a safe, non-invasive, and non-thermal modality that is based on a strong body of research dating back to the 1960.It involved in treating several conditions, the mechanisms of action involve the stimulation of mitochondria by the absorption of photons in cytochrome c oxidase, resulting in increased adenosine triphosphate production, reduced oxidative stress, anti-inflammatory effects, and increased focal cerebral blood flow

ELIGIBILITY:
Inclusion Criteria:

* Sixty elderly patients aged from 65-75 y
* Body mass index (BMI) ranged from 30 to 34.9 kg/m2
* Mild cognitive dysfunction (Montreal cognitive assessment scores from 19-25
* Anemic
* The time between their diagnoses and participation in the study ranged from 6 months to 2 years

Exclusion Criteria:

* Moderate to severe cognitive impairment
* History of neurological disease ,stroke or Cardiovascular disease
* History of nasal bleeding or fracture
* Known photo-sensitivity disorder
* Current active cancer or within one year of cancer treatment or remission
* Serious mental health illness that in the opinion of the investigator would preclude the subject from study participation
* Active infection, wound or other external trauma to the target area to receive the laser therapy
* Participation in a clinical study or other type of research in the past 30 days

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
change of cognitive function | 3 months
  comparison of Montreal assessment scale scores before and after the intervention It range between 0 and 30. A score of 26 or over is considered to be normal.
changes of hemoglobin level | 3 months
  comparison of hemoglobin level for those anemic elderly before and after the intervention
changes of balance | 3 months
  comparison of berg balance scale scores before and after the intervention. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function
changes of quality of life | 3 months
  comparison of quality of life for Alzheimer disease scores before and after the intervention. It comprised of 13 items (physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole) for a total score of 13-52 with higher scores indicating better quality of life

SECONDARY OUTCOMES:
changes of body mass index | 3 months
  comparison of body weight (kilogram) before and after the study in relation to height per meter square (weight and height will be combined to report BMI in kg/m^2)
changes of waist hip ratio | 3 months
  changes of waist hip ratio before and after the study

CONTACTS AND LOCATIONS:
Overall Officials: Ebtesam Nabil, doctoral, Principal Investigator — Cairo University
Locations (1):
- Cairo, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: after 2 years of study completion till 3 months after
Access Criteria: students and scientific researchers will be allowed to access
URL: http://Scholar.cu.edu.eg/p_t

REFERENCES:
- [Derived] Nagy EN, Ali AY, Behiry ME, Naguib MM, Elsayed MM. Impact of Combined Photo-Biomodulation and Aerobic Exercise on Cognitive Function and Quality-of-Life in Elderly Alzheimer Patients with Anemia: A Randomized Clinical Trial. Int J Gen Med. 2021 Jan 14;14:141-152. doi: 10.2147/IJGM.S280559. eCollection 2021. PMID 33469351